CLINICAL TRIAL: NCT01826968
Title: Phase 2 Study of the Alveolar Recruitment Maneuver in Cesarean Section
Brief Title: Alveolar Recruitment Maneuver During Cesarean Section Improves Lung Compliance
Acronym: CSRecGHPyr
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: General Hospital Of Pyrgos (Other)
Responsible Party: Principal Investigator, Diamanto Aretha, Anesthesiology Consultant Grade A, MD, Ph.D, General Hospital Of Pyrgos
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Lung Recruitment in Cesareans; GHPyrgosRECProt (Other: RECProt010113)
Record Dates: First submitted 2013-03-29; First posted 2013-04-09 (Estimated); Last update posted 2015-06-23 (Estimated); Status verified 2013-11

CONDITIONS: Decreased Lung Compliance; Hypoxia; Hypercapnia; Atelectasis; Pneumonia
Keywords: Lung recruitment, cesarean, lung compliance, atelectasis
MeSH Terms: conditions — Hypoxia; Hypercapnia; Pulmonary Atelectasis; Pneumonia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Recruitment Group (Experimental): The investigators used alveolar recruitment maneuver by increasing inspiratory pressure to 20 cmH20 and progressively increasing Positive Expiratory Pressure (PEEP) up to 45 cmH2O maximal (Ppeak) inspiratory pressure. The recruitment maneuver lasted 2 minutes. In this group PEEP was set to 8 cmH2O, after the recruitment maneuver, and was left until the end of the operation.
  Interventions: Procedure: Alveolar Recruitment maneuver
- Control Group (No Intervention): We did not used alveolar recruitment maneuver

INTERVENTIONS:
Procedure: Alveolar Recruitment maneuver — In this group and during recruitment maneuver the investigators used pressure control ventilation and increased inspiratory time to 50%. The investigators used alveolar recruitment maneuver by increasing inspiratory pressure to 20 cmH20 and progressively increasing Positive Expiratory Pressure (PEEP) up to 45 cmH2O maximal (Ppeak) inspiratory pressure. The recruitment maneuver lasted 2 minutes. After the maneuver PEEP was set to 8 cmH2O and was left until the end of the operation. After the end of the recruitment maneuver volume control ventilation was used until the end of the operation too.
  Arms: Recruitment Group

SUMMARY:
The investigators tested the hypothesis that alveolar recruitment maneuver during cesarean section and in women under general anesthesia improves lung compliance and gas exchange. The investigators applied recruitment maneuver and positive end expiratory pressure (PEEP) 8 cmH2O. The maximum alveolar pressure limit (Ppeak)was 45 cmH2O during the recruitment maneuver. The primary end point of the study is the improvement of the lung compliance measured as volume difference/pressure difference (dv/dp) or ml/cmH2O

DETAILED DESCRIPTION:
The investigators used recruitment maneuver during cesarean section and in women under general anesthesia. The primary end point of the study is the improvement of the lung compliance measured as volume difference/pressure difference (dv/dp) or ml/cmH2O after the recruitment maneuver. The investigators used 2 groups of patients. In the first group the investigators used pressure control ventilation for the recruitment maneuver. After the ventilator was switched to pressure control mode the investigators increased the inspiratory time to 50% and the inspiratory pressure above Positive End Expiratory Pressure (Ppeak) to 20 cmH2O. Then the investigators progressively increased Positive End Expiratory Pressure (PEEP) to have a peak inspiratory pressure (Ppeak) to 45 cm H2O. The whole recruitment maneuver lasts 2 minutes. After the recruitment maneuver the investigators used volume control ventilation again (with the baseline settings)and PEEP step wised decreased to 8 cmH20but. PEEP (8cmH2O) was left until the end of the operation. In the second group the investigators did not used lung recruitment maneuver at all. In both groups lung compliance was measured (dynamic and static)as dv/dp (ml/cmH2O). Measures were assessed 1 minute after delivery (but before recruitment), 3 minutes after recruitment (first group) at 10 and at 20 minutes after recruitment. The investigators also measured Ppeak (cmH2O) and Pplateau (cmH2O)inspiratory pressures , blood pressure (mmHG), beats per minute, oxygen saturation, end-tidal CO2 according to the above time frame, blood Gases before and 3 minutes after recruitment etc.

ELIGIBILITY:
Inclusion Criteria:

* general anesthesia,
* hemodynamically stable

Exclusion Criteria:

* intracranial hypertension,
* pulmonary hypertension,
* low blood pressure (MBP<80 mmHg),
* Heart rate > 100 beats/min,
* patient refusal

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2013-01; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Lung Compliance change measured as volume difference/pressure difference (dv/dp) or ml/cmH2O is being assessed | Before recruitment, 3 minutes after recruitment, 10 minutes after recruitment and 20 minutes after recruitment

SECONDARY OUTCOMES:
Oxygenation change is being assessed measured as PO2 (mmHg) and O2 Saturation (SPO2) | Before recruitment and 20 minutes after recruitment
Gas exchange change is being assessed measured as PCO2 (mmHg) and PH. | Before recruitment and at 20 minutes after recruitment
Pulmonary complications | up to 72 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Diamanto Aretha, MD, Principal Investigator — General Hospital of Pyrgos, Sintriada, Pyrgos, Greece
Locations (1):
- General Hospital of Pyrgos, Pýrgos, Hlia, Greece

REFERENCES:
- [Background] Valenza F, Chevallard G, Fossali T, Salice V, Pizzocri M, Gattinoni L. Management of mechanical ventilation during laparoscopic surgery. Best Pract Res Clin Anaesthesiol. 2010 Jun;24(2):227-41. doi: 10.1016/j.bpa.2010.02.002. PMID 20608559
- [Background] Strang CM, Hachenberg T, Freden F, Hedenstierna G. Development of atelectasis and arterial to end-tidal PCO2-difference in a porcine model of pneumoperitoneum. Br J Anaesth. 2009 Aug;103(2):298-303. doi: 10.1093/bja/aep102. Epub 2009 May 13. PMID 19443420
- [Background] Hedenstierna G, Edmark L. The effects of anesthesia and muscle paralysis on the respiratory system. Intensive Care Med. 2005 Oct;31(10):1327-35. doi: 10.1007/s00134-005-2761-7. Epub 2005 Aug 16. PMID 16132894
- [Background] Cinnella G, Grasso S, Spadaro S, Rauseo M, Mirabella L, Salatto P, De Capraris A, Nappi L, Greco P, Dambrosio M. Effects of recruitment maneuver and positive end-expiratory pressure on respiratory mechanics and transpulmonary pressure during laparoscopic surgery. Anesthesiology. 2013 Jan;118(1):114-22. doi: 10.1097/ALN.0b013e3182746a10. PMID 23196259